CLINICAL TRIAL: NCT02305849
Title: Phase 3 Study of ASP015K - A Randomized, Double-blind, Placebo-controlled Confirmatory Study of the Efficacy and Safety of ASP015K in Patients With Rheumatoid Arthritis Who Had an Inadequate Response to MTX
Brief Title: A Study to Evaluate Efficacy and Safety of ASP015K in Patients With Rheumatoid Arthritis (RA) Who Had an Inadequate Response to Methotrexate (MTX) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-RAJ4
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: ASP015K; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Peficitinib 100 mg (Experimental): Participants received 100 mg tablet of peficitinib orally once daily in combination with MTX for a period of 52 weeks.
  Interventions: Drug: Peficitinib; Drug: Methotrexate
- Peficitinib 150 mg (Experimental): Participants received 150 mg tablet of peficitinib orally once daily in combination with MTX for a period of 52 weeks.
  Interventions: Drug: Peficitinib; Drug: Methotrexate
- Placebo (Placebo Comparator): Participants who received placebo matching to peficitinib 100 mg or 150 mg orally once daily in combination with MTX until week 12 or 28 were switched to receive 100 mg or 150 mg tablet of peficitinib orally once daily in combination with MTX from week 12 or 28 to week 52.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Peficitinib — oral tablet
  Other Names: ASP015K
  Arms: Peficitinib 100 mg; Peficitinib 150 mg
Drug: Placebo — oral tablet
  Arms: Placebo
Drug: Methotrexate — Oral tablet/capsule

SUMMARY:
The objective of this study was to verify the efficacy of ASP015K versus placebo administrated in combination with methotrexate (MTX) over placebo in terms of efficacy in participants with rheumatoid arthritis (RA) who had an inadequate response to MTX

DETAILED DESCRIPTION:
This study was a multi-center, randomized, placebo-controlled, double-blind, parallel-group, confirmatory study to evaluate the efficacy and safety of ASP015K (100 and 150 mg/day) administered in combination with MTX in participants with RA who had an inadequate response to MTX.

Participants orally received ASP015K 100 mg, ASP015K 150 mg or placebo once daily (QD) in combination with MTX after breakfast for 52 weeks.

At Week 12, inadequate responders in the placebo group, as determined by a < 20% improvement from baseline (i.e., treatment initiation day) in tender or painful joint count (TJC) and swollen joint count (SJC), were switched to either ASP015K 100 mg or ASP015K 150 mg, and the dosage was maintained until the end of treatment (EOT). In addition, participants who received placebo at Week 28 were switched to either ASP015K 100 mg or ASP015K 150 mg, and the dosage was maintained until the EOT.

The ASP015K dose that was started for placebo group participants at Week 12 or Week 28 was randomly chosen at baseline. The dose was switched under the blinded condition.

Participants who completed this study were eligible for participation in the open-label extension study (015K-CL-RAJ2). Participants made a follow-up visit after the week 52 visit if they did not enroll into the extension study on the day of the week 52 visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject has RA of < 10 years duration at baseline that was diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria
* Subject who did not receive the following drugs, or received the drugs with stable dosage for at least 28 days prior to the baseline (start of treatment) for RA treatment:

  * Non-steroidal anti-inflammatory drugs (NSAIDs; excluding topical formulations with a local action), oral morphine or equivalent opioid analgesics (≤ 30 mg/day), acetaminophen, or oral corticosteroids (≤ 10 mg/day in prednisolone equivalent)
* At screening subject has active RA as evidenced by both of the following:

  * ≥ 6 tender/painful joints (using 68-joint assessment)
  * ≥ 6 swollen joints (using 66-joint assessment)
* CRP (latex agglutination test) of ≥ 1.00 mg/dL at screening.
* Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II or, III at screening
* Inadequate responders to MTX which was continuously administered for at least 90 days prior to screening and MTX ≥ 8 mg/week for at least 28 days prior to baseline. However, inadequate responder to MTX < 8 mg/week is eligible if intolerance precludes dose increase and defined as MTX-IR
* Subject is able to continue stable dose of MTX (a maximum of 16 mg/week) from at least 28 days prior to screening until the end of treatment
* Subject has bone erosion at the joint (as evidenced by x-rays of hands and feet) assessed in mTSS and any of the following apply at screening. Bone erosion may be evidenced by x-rays within 90 days prior to baseline.

  * Positive anti-CCP antibody: ≥ 4.5 U/mL
  * Positive rheumatoid factor: > 15 IU/mL

Exclusion Criteria:

* Subject has received a biologic DMARD within the specified period
* Inadequate responders to biologic DMARD as determined by investigator/sub-investigator
* Subject has received intra-articular, intravenous, intramuscular or endorectal (excluding suppositories for anal diseases) corticosteroid within 28 days prior to baseline
* Subject has participated in any study of ASP015K and has received ASP015K or placebo
* Subject has received other investigational drugs within 90 days or within 5 half-lives, whichever is longer, prior to baseline
* Subject has received plasma exchange therapy within 60 days prior to baseline
* Subject has undergone joint drainage, has received local anesthesia and nerve block, or has received articular cartilage protectant at the assessed joint within 28 days prior to baseline
* Subject has undergone surgery and has residual effects in the assessed joints at the discretion of investigator/sub-investigator, or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints at the discretion of investigator/sub-investigator
* A diagnosis of inflammatory arthritis (psoriatic arthritis, ankylosing spondylitis, SLE, sarcoidosis, etc.) other than RA
* Any of the following laboratory values at screening:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count < 1000/μL
  * Absolute lymphocyte count < 800/μL
  * Platelet count < 75000/μL
  * ALT ≥ 2 ×ULN
  * AST ≥ 2 × ULN
  * Total bilirubin (TBL) ≥ 1.5 × ULN
  * Estimated GFR ≤ 40 mL/min as measured by the MDRD method
  * β-D-glucan ≥ 11 pg/mL
  * Positive HBs antigen, HBc antibody, HBs antibody or HBV-DNA quantitation (However, subject with negative HBs antigen and HBV-DNA quantitation, and positive HBc antibody and/or HBs antibody is eligible if HBV-DNA is monitored by HBV-DNA quantitation at every scheduled visit after initiation of study drug administration.)
  * Positive HCV antibody
* Subject has a history of or concurrent active tuberculosis (TB)
* Subject has a history of or concurrent interstitial pneumonia and investigator/sub-investigator judges that it is inappropriate for the subject to participate in this study
* Subject has a history of or concurrent malignant tumor (except for successfully treated basal cell carcinoma)
* Subject has received live or live attenuated virus vaccination within 56 days prior to baseline. (Inactivated vaccines including influenza and pneumococcal vaccines are allowed.)
* Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA (excluding Sjogren's syndrome and chronic thyroiditis), or any ongoing illness which would make the subject unsuitable for the study as determined by the investigator/sub-investigator
* Subject has a history of clinically significant allergy. (Clinically significant allergy includes allergies such as systemic urticaria induced by specific antigens and drugs, anaphylaxis, and allergy associated with shock necessitating hospitalized treatment.)
* Subject has concurrent cardiac failure, defined as NYHA classification Class III or higher, or a history of it
* Subject has concurrent prolonged QT syndrome or a history of it. Subject has prolonged QT interval (defined as QTc ≥ 500 msec. Subject has QTc ≥ 500 msec at retest will be excluded) at screening
* Subject has a history of positive HIV infection
* Subject has congenital short QT syndrome or a history of it. Subject has shortened QT interval (defined as QTc < 330 msec. Subject has QTc < 330 msec at retest will be excluded) at screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (146):
- Japan (146):
  - JP00037, Nagoya, Aichi-ken
  - JP00109, Nagoya, Aichi-ken
  - JP00130, Nagoya, Aichi-ken
  - JP00175, Nagoya, Aichi-ken
  - JP00066, Okazaki, Aichi-ken
  - JP00108, Toyohashi, Aichi-ken
  - JP00170, Toyohashi, Aichi-ken
  - JP00156, Toyota, Aichi-ken
  - JP00068, Yatomi, Aichi-ken
  - JP00180, Asahi, Chiba
  - JP00166, Funabashi, Chiba
  - JP00115, Narashino, Chiba
  - JP00138, Yotsukaidō, Chiba
  - JP00120, Iizuka, Fukuoka
  - JP00110, Kasuga, Fukuoka
  - JP00040, Kitakyushu, Fukuoka
  - JP00119, Kitakyushu, Fukuoka
  - JP00071, Kurume, Fukuoka
  - JP00106, Kurume, Fukuoka
  - JP00033, Takasaki, Gunma
  - JP00163, Higashihiroshima, Hiroshima
  - JP00124, Tomakomai, Hokaido
  - JP00026, Asahikawa, Hokkaido
  - JP00090, Hakodate, Hokkaido
  - JP00172, Kitami, Hokkaido
  - JP00125, Kushiro, Hokkaido
  - JP00001, Sapporo, Hokkaido
  - JP00002, Sapporo, Hokkaido
  - JP00003, Sapporo, Hokkaido
  - JP00038, Sapporo, Hokkaido
  - JP00114, Sapporo, Hokkaido
  - JP00056, Akashi, Hyōgo
  - JP00069, Himeji, Hyōgo
  - JP00136, Itami, Hyōgo
  - JP00113, Kakogawa, Hyōgo
  - JP00041, Katō, Hyōgo
  - JP00042, Kobe, Hyōgo
  - JP00092, Kobe, Hyōgo
  - JP00154, Kobe, Hyōgo
  - JP00171, Kobe, Hyōgo
  - JP00117, Nishinomiya, Hyōgo
  - JP00107, Hitachi, Ibaraki
  - JP00181, Hitachi-Naka, Ibaraki
  - JP00073, Koga, Ibaraki
  - JP00054, Mito, Ibaraki
  - JP00039, Tsukuba, Ibaraki
  - JP00179, Komatsu, Ishikawa-ken
  - JP00049, Morioka, Iwate
  - JP00088, Kida, Kagawa-ken
  - JP00084, Isehara, Kanagawa
  - JP00048, Kawasaki, Kanagawa
  - JP00058, Kawasaki, Kanagawa
  - JP00141, Sagamihara, Kanagawa
  - JP00096, Yokohama, Kanagawa
  - JP00045, Zushi, Kanagawa
  - JP00019, Kōshi, Kumamoto
  - JP00057, Tamana, Kumamoto
  - JP00168, Yokkaichi, Mie-ken
  - JP00169, Ōsaki, Miyagi
  - JP00004, Sendai, Miyagi
  - JP00036, Sendai, Miyagi
  - JP00105, Sendai, Miyagi
  - JP00151, Sendai, Miyagi
  - JP00050, Hyūga, Miyazaki
  - JP00129, Matsumoto, Nagano
  - JP00162, Isehaya, Nagasaki
  - JP00101, Ōmura, Nagasaki
  - JP00103, Ōmura, Nagasaki
  - JP00153, Sasebo, Nagasaki
  - JP00094, Kashihara, Nara
  - JP00025, Nagaoka, Niigata
  - JP00144, Shibata, Niigata
  - JP00064, Beppu, Oita Prefecture
  - JP00051, Setouchi, Okayama-ken
  - JP00011, Hannan, Osaka
  - JP00134, Higashiosaka, Osaka
  - JP00178, Hirakata, Osaka
  - JP00078, Kawachi-Nagano, Osaka
  - JP00137, Sakai, Osaka
  - JP00070, Suita, Osaka
  - JP00146, Suita, Osaka
  - JP00061, Toyonaka, Osaka
  - JP00075, Ureshino, Saga-ken
  - JP00126, Gyōda, Saitama
  - JP00007, Hiki, Saitama
  - JP00060, Kawagoe, Saitama
  - JP00161, Kawagoe, Saitama
  - JP00062, Kawaguchi, Saitama
  - JP00052, Sayama, Saitama
  - JP00008, Tokorozawa, Saitama
  - JP00133, Kakegawa, Shizuoka
  - JP00077, Kanuma, Tochigi
  - JP00145, Shimotsuke, Tochigi
  - JP00024, Bunkyo, Tokyo
  - JP00143, Bunkyo, Tokyo
  - JP00149, Bunkyo, Tokyo
  - JP00152, Bunkyo, Tokyo
  - JP00099, Chiyoda City, Tokyo
  - JP00142, Chūō, Tokyo
  - JP00063, Hachiōji, Tokyo
  - JP00053, Kiyose, Tokyo
  - JP00072, Meguro City, Tokyo
  - JP00148, Ōta-ku, Tokyo
  - JP00081, Shibuya City, Tokyo
  - JP00010, Takaoka, Toyama
  - JP00155, Nishimuro, Wakayama
  - JP00104, Shimonoseki, Yamaguchi
  - JP00047, Shūnan, Yamaguchi
  - JP00176, Fukui
  - JP00018, Fukuoka
  - JP00020, Fukuoka
  - JP00035, Fukuoka
  - JP00059, Fukuoka
  - JP00067, Fukuoka
  - JP00076, Fukuoka
  - JP00131, Fukuoka
  - JP00164, Fukuoka
  - JP00165, Fukushima
  - JP00013, Hiroshima
  - JP00014, Hiroshima
  - JP00016, Hiroshima
  - JP00055, Hiroshima
  - JP00074, Kagoshima
  - JP00167, Kagoshima
  - JP00093, Kochi
  - JP00022, Kumamoto
  - JP00046, Kumamoto
  - JP00085, Kyoto
  - JP00123, Kyoto
  - JP00160, Kyoto
  - JP00023, Miyagi
  - JP00122, Miyazaki
  - JP00080, Nagano
  - JP00174, Nagano
  - JP00098, Nagasaki
  - JP00112, Nagasaki
  - JP00147, Nagasaki
  - JP00118, Okayama
  - JP00150, Osaka
  - JP00157, Osaka
  - JP00177, Osaka
  - JP00017, Ōita
  - JP00044, Shizuoka
  - JP00089, Shizuoka
  - JP00135, Shizuoka
  - JP00139, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tanaka Y, Takeuchi T, Kato D, Kaneko Y, Fukuda M, Izutsu H, Rokuda M, van der Heijde D. Post hoc analysis of clinical characteristics of patients with radiographic progression in a Japanese phase 3 trial of peficitinib and methotrexate treatment (RAJ4). Mod Rheumatol. 2023 Jan 3;33(1):73-80. doi: 10.1093/mr/roac021. PMID 35267027
- [Derived] Tanaka Y, Takeuchi T, Izutsu H, Kaneko Y, Kato D, Fukuda M, Rokuda M, Schultz NM. Patient- and physician-reported outcomes from two phase 3 randomized studies (RAJ3 and RAJ4) of peficitinib (ASP015K) in Asian patients with rheumatoid arthritis. Arthritis Res Ther. 2021 Aug 24;23(1):221. doi: 10.1186/s13075-021-02590-z. PMID 34429152
- [Derived] Toyoshima J, Kaibara A, Shibata M, Kaneko Y, Izutsu H, Nishimura T. Exposure-response modeling of peficitinib efficacy in patients with rheumatoid arthritis. Pharmacol Res Perspect. 2021 May;9(3):e00744. doi: 10.1002/prp2.744. PMID 33929089
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028
- [Derived] Takeuchi T, Tanaka Y, Tanaka S, Kawakami A, Iwasaki M, Katayama K, Rokuda M, Izutsu H, Ushijima S, Kaneko Y, Shiomi T, Yamada E, van der Heijde D. Efficacy and safety of peficitinib (ASP015K) in patients with rheumatoid arthritis and an inadequate response to methotrexate: results of a phase III randomised, double-blind, placebo-controlled trial (RAJ4) in Japan. Ann Rheum Dis. 2019 Oct;78(10):1305-1319. doi: 10.1136/annrheumdis-2019-215164. Epub 2019 Jul 26. PMID 31350269
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with rheumatoid arthritis (RA) who had an inadequate response to methotrexate (MTX) were enrolled in this study.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to peficitinib 100 milligram (mg), 150 mg or placebo groups in combination with MTX at baseline. At week 12 or 28, participants in the placebo group were switched to receive either peficitinib at a dose of 100 mg or 150 mg, which was determined in advance randomly.
Groups:
- Placebo / Peficitinib 100 mg: Participants who received placebo matching to peficitinib 100 mg orally once daily in combination with MTX until week 12 or 28 were switched to receive 100 mg tablet of peficitinib orally once daily in combination with MTX from week 12 or 28 to week 52.
- Placebo / Peficitinib 150 mg: Participants who received placebo matching to peficitinib 150 mg orally once daily in combination with MTX until week 12 or 28 were switched to receive 150 mg tablet of peficitinib orally once daily in combination with MTX from week 12 or 28 to week 52.
Period: Overall Study
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg
Started | 175 | 174 | 85 | 85
Completed | 148 | 146 | 67 | 66
Not Completed | 27 | 28 | 18 | 19
Not completed — Adverse Event | 10 | 12 | 7 | 3
Not completed — Lack of Efficacy | 10 | 6 | 3 | 9
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 1 | 1
Not completed — Lab data met discontinuation criteria | 0 | 1 | 2 | 1
Not completed — Miscellaneous | 1 | 2 | 4 | 1
Not completed — Not fulfill eligibility criteria | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) was defined as all participants who received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo | Total
Number analyzed (Participants) | 174 | 174 | 170 | 518
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (10.8) | 56.2 (11.6) | 55.3 (12.1) | 56.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 125 | 121 | 364
  Male | 56 | 49 | 49 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 174 | 174 | 170 | 518
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] — Higher CRP indicates greater disease activity. Population: Full analysis set (FAS) included all participants who were randomized and received at least one dose of the study drug. Here, Number of participants analyzed signifies participants with available data.
  milligram/deciliter (mg/dL)
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 2.432 (2.076) | 2.524 (2.183) | 2.622 (2.146) | 2.525 (2.132)
Erosion Score [Mean (Standard Deviation); unit: units on a scale] — The joint erosion score was a summary of erosion severity in 32 joints of the hands and 12 joints of the feet. Each joint in the hand is scored from 0-5 and each joint in the foot is scored from 0-10. The score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet. By summing these score, the range of total erosion score is 0-280. Higher erosion score indicates greater disease activity. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 173 | 174 | 169 | 516
    (all) | 10.34 (17.47) | 9.76 (15.93) | 11.03 (17.96) | 10.37 (17.11)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: millimeter per hour (mm/h)] — Population: FAS.
  millimeter per hour (mm/h) | 50.4 (26.2) | 51.5 (26.8) | 53.8 (26.9) | 51.9 (26.6)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — Participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 0.91 (0.65) | 1.02 (0.62) | 1.05 (0.66) | 0.99 (0.65)
Joint Space Narrowing (JSN) Score [Mean (Standard Deviation); unit: units on a scale] — JSN was defined as narrowing in joint space width over the course of the study. The JSN score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet. JSN, including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. Higher joint space narrowing score indicates greater disease activity. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 173 | 174 | 169 | 516
    (all) | 14.89 (19.47) | 15.23 (18.33) | 17.37 (20.13) | 15.82 (19.31)
Modified Total Sharp Score (mTSS) [Mean (Standard Deviation); unit: units on a scale] — mTSS was defined as the sum of joint erosion scores graded by assessing erosion severity in 44 joints and JSN scores graded by assessing narrowing of joint spaces in 42 joints. mTSS scores ranged from 0 (normal) to 448 (worst possible total score). An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 173 | 174 | 169 | 516
    (all) | 25.23 (35.5) | 25 (32.38) | 28.4 (36.28) | 26.19 (34.71)
Physician's Global Assessment of Arthritis (PGA) [Mean (Standard Deviation); unit: units on a scale] — Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm visual analog scale (VAS) where 0 = very well and 100 = very poorly. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 58.87 (19.67) | 60.86 (19.09) | 60.98 (19.59) | 60.23 (19.43)
Subject's Global Assessment of Arthritis (SGA) [Mean (Standard Deviation); unit: units on a scale] — Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 51.7 (25.25) | 55.44 (24.49) | 58.18 (23.9) | 55.07 (24.65)
Subject's Global Assessment of Arthritis Pain (SGAP) [Mean (Standard Deviation); unit: units on a scale] — The participant assessed his/her own pain severity on a visual analog scale (VAS) of 0-100 mm on the questionnaire form. Higher SGAP (100 mm VAS) scores indicated greater activity pain. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  units on a scale
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 51.12 (26.14) | 55.09 (24.89) | 56.75 (25.29) | 54.3 (25.51)
Swollen Joint Count (SJC) (66 Joints) [Mean (Standard Deviation); unit: swollen joint count] — The participants were examined for the swollen joints and the location was confirmed by the investigator who assessed the 66 joints. Higher SJC indicated greater disease activity. Population: FAS.
  swollen joint count | 12.8 (6.8) | 13.1 (6.9) | 13.6 (7) | 13.2 (6.9)
Tender Joint Count (TJC) (68 Joints) [Mean (Standard Deviation); unit: tender joint count] — The participants were examined for the tender joints and the location was confirmed by the investigator who assessed the 68 joints. Higher TJC indicated greater disease activity. Population: FAS. Here, Number of participants analyzed signifies participants with available data.
  tender joint count
    number analyzed (Participants) | 174 | 174 | 169 | 517
    (all) | 14 (8.6) | 14.5 (7.8) | 15.4 (9.4) | 14.6 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) C-Reactive Protein (CRP) Response at Week 12
Description: ACR20 response: greater than and equal to (≥) 20 percent (%) improvement in tender and swollen joint count; and ≥ 20% improvement in at least 3 of the following 5 criteria compared with baseline: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Baseline and week 12/Early termination (ET)
Population: FAS. Last observation carried forward (LOCF) was used for missing imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 170 | 174 | 174
percentage of participants | 21.8 | 58.6 | 64.4
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Closed testing procedure was used for multiplicity adjustment; Percent Difference = 36.9, 95% CI 2-sided [26.7 to 47.0] — CI was based on normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Closed testing procedure was used for multiplicity adjustment; Percent difference = 42.6, 95% CI 2-sided [32.6 to 52.6] — CI was based on normal approximation to the binomial distribution

2. Primary Outcome: Change From Baseline in mTSS at Week 28
Description: mTSS was defined as the sum of joint erosion scores graded by assessing erosion severity in 44 joints (16 per hand and 6 per feet) and JSN scores graded by assessing narrowing of joint spaces in 42 joints (15 per hand and 6 per feet). Erosion score was scored from 0 (no erosion) to 5 (complete collapse of bone) and the score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet (the maximum erosion score for a joint in the foot is 10). JSN including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change from baseline was calculated as score at week 28 (ET) minus score at baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and week 28/ET
Population: FAS. Here, Number of participants analyzed signifies participants with available data. Missing values were imputed by linear extrapolation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 153 | 164 | 164
units on a scale | 3.37 (5.46) | 1.62 (4.23) | 1.03 (2.86)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA — Closed testing procedure was used for multiplicity adjustment; Based on Rank Analysis of Covariance (RANCOVA) Model: Rank of mTSS Change = Treatment + Baseline Rank of mTSS
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA — Closed testing procedure was used for multiplicity adjustment; Based on RANCOVA Model: Rank of mTSS Change = Treatment + Baseline Rank of mTSS

3. Secondary Outcome: Percentage of Participants With an ACR20-CRP Response Through Week 52
Description: ACR20 response:≥ 20% improvement in tender and swollen joint count; and ≥ 20% improvement in at least 3 of the following 5 criteria compared with baseline: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit. EOT was defined as end of treatment i.e, either early termination or week 52.
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, number of participants analyzed signifies participants with available data.
Measure: Number; unit: percentage of participants
Groups:
- Placebo / Peficitinib 100 mg at Week 12: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 12 were switched to receive 100 mg tablet of peficitinib orally once daily in combination with MTX from week 12 to week 52.
- Placebo / Peficitinib 150 mg at Week 12: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 12 were switched to receive 150 mg tablet of peficitinib orally once daily in combination with MTX from week 12 to week 52.
- Placebo / Peficitinib 100 mg at Week 28: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 28 were switched to receive 100 mg tablet of peficitinib orally once daily in combination with MTX from week 28 to week 52.
- Placebo / Peficitinib 150 mg at Week 28: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 28 were switched to receive 150 mg tablet of peficitinib orally once daily in combination with MTX from week 28 to week 52.
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 174 | 174 | 37 | 38 | 39 | 34
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 37 | 39 | 34
  Week 4 | 38.2 | 48.2 | 8.1 | 2.7 | 38.5 | 14.7
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 8 | 51.2 | 62.0 | 10.8 | 0.0 | 33.3 | 29.4
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | 59.5 | 66.3 | 0.0 | 0.0 | 51.3 | 38.2
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | 70.5 | 77.0 | 43.2 | 51.4 | 64.1 | 58.8
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | 74.4 | 79.8 | 59.5 | 67.6 | 61.5 | 61.8
  Week 24: number analyzed (Participants) | 161 | 160 | 36 | 36 | 39 | 34
  Week 24 | 74.5 | 85.0 | 63.9 | 80.6 | 59.0 | 52.9
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | 79.1 | 83.0 | 72.2 | 83.3 | 64.1 | 64.7
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | 79.6 | 85.2 | 77.8 | 86.1 | 84.6 | 76.5
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | 78.4 | 86.5 | 80.6 | 85.7 | 78.4 | 75.8
  Week 40: number analyzed (Participants) | 152 | 153 | 35 | 34 | 36 | 33
  Week 40 | 80.9 | 86.9 | 80.0 | 88.2 | 88.9 | 78.8
  Week 44: number analyzed (Participants) | 149 | 153 | 34 | 33 | 36 | 33
  Week 44 | 79.9 | 86.9 | 76.5 | 90.9 | 88.9 | 87.9
  Week 48: number analyzed (Participants) | 148 | 151 | 33 | 33 | 35 | 33
  Week 48 | 83.8 | 89.4 | 81.8 | 90.9 | 85.7 | 90.9
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | 84.8 | 87.1 | 75.8 | 90.9 | 91.2 | 90.9
  EOT | 76.4 | 81.0 | 73.0 | 78.9 | 92.3 | 91.2

4. Secondary Outcome: Percentage of Participants With an ACR50-CRP Response at Week 12
Description: ACR50 response: ≥50% improvement in tender and swollen joint counts and 50% improvement in 3 of the following 5 criteria compared with baseline: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) C-reactive protein at each visit.
Time Frame: Baseline and week 12/ET
Population: FAS. LOCF was used for missing imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 170 | 174 | 174
percentage of participants | 7.6 | 29.9 | 46.0
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 22.2, 95% CI 2-sided [13.8 to 30.7] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 38.3, 95% CI 2-sided [29.3 to 47.3] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

5. Secondary Outcome: Percentage of Participants With an ACR50-CRP Response Through Week 52
Description: as for outcome 4
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 174 | 174 | 37 | 38 | 39 | 34
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 37 | 39 | 34
  Week 4 | 10.0 | 15.9 | 2.7 | 0.0 | 10.3 | 0.0
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 8 | 19.6 | 33.1 | 2.7 | 0.0 | 12.8 | 2.9
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | 29.8 | 48.2 | 0.0 | 0.0 | 23.1 | 5.9
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | 46.4 | 53.9 | 13.5 | 21.6 | 38.5 | 8.8
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | 51.2 | 54.6 | 35.1 | 37.8 | 35.9 | 29.4
  Week 24: number analyzed (Participants) | 161 | 160 | 36 | 36 | 39 | 34
  Week 24 | 56.5 | 60.6 | 47.2 | 52.8 | 33.3 | 29.4
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | 53.8 | 63.5 | 50.0 | 69.4 | 28.2 | 23.5
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | 59.2 | 65.8 | 52.8 | 61.1 | 56.4 | 52.9
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | 55.6 | 67.7 | 58.3 | 71.4 | 64.9 | 60.6
  Week 40: number analyzed (Participants) | 152 | 153 | 35 | 34 | 36 | 33
  Week 40 | 61.8 | 68.0 | 48.6 | 67.6 | 66.7 | 66.7
  Week 44: number analyzed (Participants) | 149 | 153 | 34 | 33 | 36 | 33
  Week 44 | 57.7 | 71.2 | 52.9 | 72.7 | 72.2 | 63.6
  Week 48: number analyzed (Participants) | 148 | 151 | 33 | 33 | 35 | 33
  Week 48 | 60.8 | 64.9 | 60.6 | 69.7 | 71.4 | 66.7
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | 66.9 | 68.0 | 63.6 | 63.6 | 67.6 | 69.7
  EOT | 60.3 | 62.6 | 62.2 | 55.3 | 69.2 | 70.6

6. Secondary Outcome: Percentage of Participants With an ACR70-CRP Response at Week 12
Description: ACR70 response: ≥ 70% improvement in tender and swollen joint counts and 70% improvement in 3 of the following 5 criteria compared with baseline: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) C-reactive protein at each visit.
Time Frame: Baseline and week 12/ET
Population: FAS. LOCF was used for missing imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 170 | 174 | 174
percentage of participants | 2.4 | 12.1 | 23.6
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 9.7, 95% CI 2-sided [3.8 to 15.6] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 21.2, 95% CI 2-sided [13.9 to 28.5] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

7. Secondary Outcome: Percentage of Participants With an ACR70-CRP Response Through Week 52
Description: as for outcome 6
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 174 | 174 | 37 | 38 | 39 | 34
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 37 | 39 | 34
  Week 4 | 1.2 | 4.1 | 0.0 | 0.0 | 2.6 | 0.0
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 8 | 7.7 | 13.9 | 0.0 | 0.0 | 2.6 | 0.0
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | 12.5 | 24.7 | 0.0 | 0.0 | 7.7 | 2.9
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | 24.1 | 32.1 | 5.4 | 2.7 | 12.8 | 2.9
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | 26.2 | 35.0 | 8.1 | 2.7 | 12.8 | 2.9
  Week 24: number analyzed (Participants) | 161 | 161 | 36 | 36 | 39 | 34
  Week 24 | 31.7 | 36.0 | 22.2 | 16.7 | 17.9 | 2.9
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | 29.1 | 42.8 | 33.3 | 38.9 | 17.9 | 8.8
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | 36.3 | 43.9 | 33.3 | 44.4 | 20.5 | 20.6
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | 34.0 | 47.1 | 33.3 | 42.9 | 13.5 | 33.3
  Week 40: number analyzed (Participants) | 152 | 153 | 35 | 34 | 36 | 33
  Week 40 | 34.9 | 41.8 | 31.4 | 38.2 | 36.1 | 33.3
  Week 44: number analyzed (Participants) | 149 | 153 | 34 | 33 | 36 | 33
  Week 44 | 38.3 | 48.4 | 41.2 | 36.4 | 38.9 | 39.4
  Week 48: number analyzed (Participants) | 148 | 151 | 33 | 33 | 35 | 33
  Week 48 | 33.8 | 49.0 | 45.5 | 42.4 | 45.7 | 39.4
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | 39.3 | 52.4 | 42.4 | 48.5 | 44.1 | 48.5
  EOT | 35.1 | 48.3 | 40.5 | 42.1 | 43.6 | 50.0

8. Secondary Outcome: Change From Baseline in mTSS at Week 52
Description: mTSS was defined as the sum of joint erosion scores graded by assessing erosion severity in 44 joints (16 per hand and 6 per feet) and JSN scores graded by assessing narrowing of joint spaces in 42 joints (15 per hand and 6 per feet). Erosion score was scored from 0 (no erosion) to 5 (complete collapse of bone) and the score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet (the maximum erosion score for a joint in the foot is 10). JSN including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change from baseline was calculated as score at week 52 (ET) minus score at baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and week 52/ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 153 | 164 | 164
units on a scale | 6.27 (10.18) | 2.12 (5.83) | 1.54 (4.11)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA — Based on RANCOVA Model: Rank of mTSS Change = Treatment + Baseline Rank of mTSS
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA — Based on RANCOVA Model: Rank of mTSS Change = Treatment + Baseline Rank of mTSS

9. Secondary Outcome: Change From Baseline in JSN Score at Week 28 and Week 52
Description: JSN was defined as narrowing in joint space width over the course of the study. The JSN score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet. JSN, including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. Higher scores indicate greater disease activity.
Time Frame: Baseline and weeks 28/ET and 52/ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 153 | 164 | 164
units on a scale
  Week 28/ET | 1.90 (3.76) | 0.99 (2.86) | 0.82 (2.39)
  Week 52/ET | 3.55 (7.01) | 1.30 (3.37) | 1.19 (3.03)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.018, RANCOVA; Based on RANCOVA Model: Rank of JSN Score Change = Treatment + Baseline Rank of JSN score
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.002, RANCOVA; Based on RANCOVA Model: Rank of JSN Score Change = Treatment + Baseline Rank of JSN score
Statistical Analysis 3: Comparison: Placebo vs Peficitinib 100 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.039, RANCOVA; Based on RANCOVA Model: Rank of JSN Score Change = Treatment + Baseline Rank of JSN Score
Statistical Analysis 4: Comparison: Placebo vs Peficitinib 150 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.006, RANCOVA; Based on RANCOVA Model: Rank of JSN Score Change = Treatment + Baseline Rank of JSN Score

10. Secondary Outcome: Change From Baseline in Erosion Score at Week 28 and Week 52
Description: The joint erosion score was a summary of erosion severity in 32 joints of the hands and 12 joints of the feet. Each joint in the hand is scored from 0-5 and each joint in the foot is scored from 0-10. The score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet. By summing these score, the range of total erosion score is 0-280. Higher erosion score indicates greater disease activity.
Time Frame: Baseline and weeks 28/ET and 52/ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 153 | 164 | 164
units on a scale
  Week 28/ET | 1.35 (3.01) | 0.63 (2.03) | 0.18 (1.10)
  Week 52/ET | 2.52 (5.58) | 0.82 (3.14) | 0.32 (1.87)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.036, RANCOVA; Based on RANCOVA Model: Rank of Erosion Score Change = Treatment + Baseline Rank of Erosion Score
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA; Based on RANCOVA Model: Rank of Erosion Score Change = Treatment + Baseline Rank of Erosion Score
Statistical Analysis 3: Comparison: Placebo vs Peficitinib 100 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p = 0.013, RANCOVA; Based on RANCOVA Model: Rank of Erosion Score Change = Treatment + Baseline Rank of Erosion Score
Statistical Analysis 4: Comparison: Placebo vs Peficitinib 150 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, RANCOVA; Based on RANCOVA Model: Rank of Erosion Score Change = Treatment + Baseline Rank of Erosion Score

11. Secondary Outcome: Percentage of Participants Achieving Change From Baseline in mTSS <= 0.5 at Week 28 and Week 52
Description: mTSS was defined as the sum of joint erosion scores graded by assessing erosion severity in 44 joints (16 per hand and 6 per feet) and JSN scores graded by assessing narrowing of joint spaces in 42 joints (15 per hand and 6 per feet). Erosion score was scored from 0 (no erosion) to 5 (complete collapse of bone) and the score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet (the maximum erosion score for a joint in the foot is 10). JSN including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. mTSS scores ranged from 0 (normal) to 448 (worst possible total score). An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and week 28/ET and 52/ET
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 153 | 164 | 164
percentage of participants
  Week 28/ET | 45.8 | 67.1 | 72.6
  Week 52/ET | 42.5 | 64.0 | 68.9
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 21.3, 95% CI 2-sided [10.0 to 32.6] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Week 28/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 26.8, 95% CI 2-sided [15.7 to 37.9] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 3: Comparison: Placebo vs Peficitinib 100 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 21.5, 95% CI 2-sided [10.2 to 32.9] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 4: Comparison: Placebo vs Peficitinib 150 mg; Week 52/ET: Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 26.4, 95% CI 2-sided [15.2 to 37.6] — CI was based on normal approximation to the binomial distribution (continuity corrected)

12. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28-CRP at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: Baseline and week 12/ET
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -0.51 (1.10) | -1.70 (1.20) | -2.09 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA (analysis of covariance) Model: DAS28 Change = Treatment + Baseline DAS28; LS Mean difference = -1.21, 95% CI 2-sided [-1.46 to -0.97], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: DAS28 Change = Treatment + Baseline DAS28; LS Mean difference = -1.59, 95% CI 2-sided [-1.85 to -1.33], Standard Error of Mean 0.13

13. Secondary Outcome: Change From Baseline in DAS28-CRP Through Week 52
Description: as for outcome 12
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, number of participants analyzed signifies participants with available data. LOCF was used for missing imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 172 | 171 | 37 | 37 | 39 | 34
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 37 | 39 | 34
  Week 4 | -1.11 (0.81) | -1.39 (0.98) | -0.28 (0.67) | -0.30 (0.56) | -0.82 (1.09) | -0.74 (0.62)
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 8 | -1.48 (1.00) | -1.87 (1.16) | -0.21 (0.86) | -0.10 (0.63) | -0.94 (0.97) | -0.90 (0.65)
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | -1.72 (1.19) | -2.15 (1.29) | 0.24 (0.75) | 0.27 (0.60) | -1.34 (1.00) | -1.20 (0.66)
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | -2.01 (1.18) | -2.40 (1.30) | -1.11 (1.15) | -1.37 (1.18) | -1.37 (1.35) | -1.31 (0.74)
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | -2.21 (1.24) | -2.53 (1.29) | -1.69 (1.22) | -1.76 (1.24) | -1.38 (1.19) | -1.48 (0.78)
  Week 24: number analyzed (Participants) | 161 | 160 | 36 | 36 | 39 | 34
  Week 24 | -2.40 (1.21) | -2.71 (1.18) | -2.01 (1.26) | -2.26 (1.07) | -1.41 (1.32) | -1.64 (0.92)
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | -2.42 (1.21) | -2.70 (1.25) | -2.24 (1.11) | -2.51 (1.13) | -1.53 (1.39) | -1.71 (0.97)
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | -2.50 (1.18) | -2.77 (1.19) | -2.49 (1.24) | -2.72 (1.27) | -2.18 (1.27) | -2.47 (0.89)
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | -2.55 (1.12) | -2.83 (1.20) | -2.49 (1.14) | -2.70 (1.22) | -2.22 (1.23) | -2.57 (0.89)
  Week 40: number analyzed (Participants) | 152 | 153 | 35 | 34 | 36 | 33
  Week 40 | -2.66 (1.16) | -2.86 (1.14) | -2.66 (1.24) | -2.72 (1.13) | -2.62 (1.05) | -2.73 (0.93)
  Week 44: number analyzed (Participants) | 149 | 153 | 34 | 33 | 36 | 33
  Week 44 | -2.65 (1.13) | -2.88 (1.15) | -2.68 (1.23) | -2.72 (1.19) | -2.63 (1.35) | -2.87 (0.89)
  Week 48: number analyzed (Participants) | 148 | 151 | 33 | 33 | 35 | 33
  Week 48 | -2.62 (1.15) | -2.92 (1.14) | -2.86 (1.26) | -2.90 (1.18) | -2.66 (1.49) | -2.96 (0.97)
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | -2.67 (1.19) | -2.96 (1.24) | -2.80 (1.46) | -2.74 (1.13) | -2.70 (1.32) | -2.89 (0.92)
  EOT | -2.43 (1.37) | -2.76 (1.40) | -2.61 (1.62) | -2.52 (1.25) | -2.72 (1.26) | -2.87 (0.92)

14. Secondary Outcome: Change From Baseline in DAS28-ESR at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: Baseline and week 12/ET
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 170
units on a scale | -0.51 (1.11) | -1.66 (1.22) | -2.12 (1.36)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: DAS28 Change = Treatment + Baseline DAS28; LS Mean difference = -1.19, 95% CI 2-sided [-1.44 to -0.94], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: DAS28 Change = Treatment + Baseline DAS28; LS Mean difference = -1.63, 95% CI 2-sided [-1.89 to -1.36], Standard Error of Mean 0.13

15. Secondary Outcome: Change From Baseline in DAS28-ESR Score Through Week 52
Description: as for outcome 14
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 172 | 170 | 37 | 37 | 39 | 34
units on a scale
  Week 4: number analyzed (Participants) | 170 | 169 | 37 | 37 | 39 | 34
  Week 4 | -1.07 (0.83) | -1.37 (1.02) | -0.26 (0.66) | -0.26 (0.59) | -0.87 (1.08) | -0.67 (0.64)
  Week 8: number analyzed (Participants) | 168 | 165 | 37 | 37 | 39 | 34
  Week 8 | -1.47 (1.06) | -1.88 (1.18) | -0.24 (0.88) | -0.12 (0.64) | -1.00 (0.93) | -0.85 (0.76)
  Week 12: number analyzed (Participants) | 168 | 165 | 37 | 37 | 39 | 34
  Week 12 | -1.68 (1.21) | -2.18 (1.32) | 0.24 (0.76) | 0.25 (0.59) | -1.40 (0.99) | -1.10 (0.76)
  Week 16: number analyzed (Participants) | 166 | 164 | 37 | 37 | 39 | 34
  Week 16 | -1.98 (1.22) | -2.46 (1.32) | -1.01 (1.14) | -1.38 (1.21) | -1.47 (1.39) | -1.21 (0.82)
  Week 20: number analyzed (Participants) | 164 | 162 | 37 | 37 | 39 | 34
  Week 20 | -2.23 (1.27) | -2.60 (1.35) | -1.61 (1.23) | -1.78 (1.26) | -1.45 (1.19) | -1.37 (0.81)
  Week 24: number analyzed (Participants) | 161 | 159 | 36 | 36 | 39 | 34
  Week 24 | -2.43 (1.28) | -2.78 (1.25) | -1.94 (1.24) | -2.24 (1.16) | -1.47 (1.31) | -1.56 (0.99)
  Week 28: number analyzed (Participants) | 158 | 158 | 36 | 36 | 39 | 34
  Week 28 | -2.47 (1.31) | -2.79 (1.29) | -2.11 (1.16) | -2.48 (1.15) | -1.63 (1.41) | -1.62 (1.07)
  Week 32: number analyzed (Participants) | 157 | 154 | 36 | 36 | 39 | 34
  Week 32 | -2.56 (1.31) | -2.87 (1.27) | -2.39 (1.26) | -2.68 (1.30) | -2.27 (1.34) | -2.37 (1.05)
  Week 36: number analyzed (Participants) | 153 | 154 | 36 | 35 | 37 | 33
  Week 36 | -2.59 (1.23) | -2.91 (1.25) | -2.45 (1.20) | -2.71 (1.20) | -2.38 (1.29) | -2.54 (1.02)
  Week 40: number analyzed (Participants) | 151 | 151 | 35 | 34 | 36 | 33
  Week 40 | -2.70 (1.22) | -2.96 (1.20) | -2.60 (1.34) | -2.78 (1.11) | -2.71 (1.16) | -2.68 (0.96)
  Week 44: number analyzed (Participants) | 147 | 152 | 34 | 33 | 36 | 33
  Week 44 | -2.71 (1.19) | -3.00 (1.25) | -2.63 (1.25) | -2.76 (1.25) | -2.74 (1.43) | -2.78 (1.04)
  Week 48: number analyzed (Participants) | 147 | 150 | 33 | 33 | 35 | 33
  Week 48 | -2.64 (1.20) | -3.01 (1.22) | -2.80 (1.36) | -2.88 (1.23) | -2.72 (1.58) | -2.93 (1.06)
  Week 52: number analyzed (Participants) | 145 | 146 | 33 | 33 | 34 | 33
  Week 52 | -2.70 (1.27) | -3.07 (1.28) | -2.77 (1.54) | -2.78 (1.24) | -2.79 (1.33) | -2.85 (1.08)
  EOT | -2.47 (1.43) | -2.86 (1.44) | -2.60 (1.69) | -2.56 (1.34) | -2.80 (1.27) | -2.82 (1.08)

16. Secondary Outcome: Change From Baseline in TJC (68 Joints) at Week 12
Description: The participants were examined for the tender joints and the location was confirmed by the investigator who assessed the following 68 joints which included temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8). Higher TJC indicated greater disease activity.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
tender joint count | -2.1 (8.2) | -6.9 (8.6) | -9.1 (8.0)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: TJC68 Change = Treatment + Baseline TJC68; LS Mean difference = -5.2, 95% CI [-6.9 to -3.5], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: TJC68 Change = Treatment + Baseline TJC68; LS Mean difference = -7.2, 95% CI 2-sided [-8.9 to -5.6], Standard Error of Mean 0.8

17. Secondary Outcome: Change From Baseline in TJC (68 Joints) Through Week 52
Description: as for outcome 16
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data. Only peficitinib 100mg and 150 mg arms are analyzed for this outcome measure, as planned.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
tender joint count
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -5.1 (5.8) | -6.3 (6.9)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -6.8 (7.2) | -8.3 (7.3)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -7.1 (8.6) | -9.3 (7.7)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -8.1 (7.8) | -10.5 (7.4)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -9.1 (7.9) | -10.8 (8.0)
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | -9.9 (7.5) | -11.3 (7.6)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -9.6 (7.4) | -11.4 (7.8)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -9.7 (7.2) | -12.1 (7.6)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -10.4 (7.6) | -11.8 (7.7)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -10.8 (7.2) | -11.9 (8.2)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -10.6 (7.4) | -12.1 (7.8)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -10.5 (7.1) | -12.1 (7.7)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -10.8 (7.4) | -11.9 (8.6)
  EOT | -9.8 (7.8) | -11.2 (8.8)

18. Secondary Outcome: Change From Baseline in SJC (66 Joints) at Week 12
Description: The participants were examined for the swollen joints and the location was confirmed by the investigator who assessed the following 66 joints which included temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8). Higher SJC indicated greater disease activity.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
swollen joint count | -2.2 (6.6) | -5.9 (6.7) | -7.6 (6.1)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SJC66 Change = Treatment + Baseline SJC66; LS Mean difference = -3.9, 95% CI 2-sided [-5.3 to -2.6], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SJC66 Change = Treatment + Baseline SJC66; LS Mean difference = -5.6, 95% CI 2-sided [-6.9 to -4.3], Standard Error of Mean 0.6

19. Secondary Outcome: Change From Baseline in SJC (66 Joints) Through Week 52
Description: as for outcome 18
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data. Only peficitinib 100 mg and 150 mg arms are analyzed for this outcome measure, as planned.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
swollen joint count
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -4.3 (4.5) | -5.3 (5.6)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -5.6 (5.5) | -7.1 (5.5)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -6.0 (6.7) | -7.8 (5.9)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -7.5 (6.2) | -8.9 (6.0)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -8.1 (6.1) | -9.2 (5.7)
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | -8.8 (6.4) | -9.9 (5.6)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -8.8 (6.2) | -9.8 (5.7)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -9.0 (6.2) | -10.3 (5.8)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -9.0 (6.1) | -10.5 (5.9)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -9.4 (6.1) | -10.7 (6.1)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -9.4 (6.1) | -10.8 (6.4)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -9.2 (6.2) | -11.0 (6.3)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -9.6 (6.2) | -11.0 (6.1)
  EOT | -8.8 (6.6) | -10.3 (6.4)

20. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score < 2.6 at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. If the DAS28 score was less than 2.6, the participant was considered to be in DAS28 remission.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 7.7 | 31.4 | 35.1
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 23.7, 95% CI 2-sided [15.1 to 32.3] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 27.4, 95% CI 2-sided [18.6 to 36.2] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

21. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score < 2.6 Through Week 52
Description: as for outcome 20
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 172 | 171 | 37 | 38 | 39 | 34
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 38 | 39 | 34
  Week 4 | 11.2 | 14.7 | 0.0 | 0.0 | 15.4 | 5.9
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 38 | 39 | 34
  Week 8 | 19.0 | 21.7 | 0.0 | 0.0 | 10.3 | 11.8
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | 31.0 | 36.1 | 0.0 | 0.0 | 20.5 | 11.8
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | 39.2 | 43.0 | 8.1 | 13.5 | 20.5 | 8.8
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | 45.7 | 52.1 | 21.6 | 16.2 | 17.9 | 29.4
  Week 24: number analyzed (Participants) | 161 | 160 | 36 | 36 | 39 | 34
  Week 24 | 51.6 | 56.9 | 27.8 | 33.3 | 20.5 | 32.4
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | 51.9 | 52.8 | 30.6 | 38.9 | 25.6 | 26.5
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | 54.1 | 52.9 | 44.4 | 50.0 | 30.8 | 44.1
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | 53.6 | 53.5 | 50.0 | 48.6 | 35.1 | 54.5
  Week 40: number analyzed (Participants) | 152 | 153 | 35 | 34 | 36 | 33
  Week 40 | 59.9 | 58.8 | 42.9 | 50.0 | 61.1 | 54.5
  Week 44: number analyzed (Participants) | 149 | 153 | 34 | 33 | 36 | 33
  Week 44 | 57.0 | 55.6 | 50.0 | 42.4 | 55.6 | 57.6
  Week 48: number analyzed (Participants) | 148 | 151 | 33 | 33 | 35 | 33
  Week 48 | 56.1 | 60.3 | 54.5 | 54.5 | 62.9 | 66.7
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | 60.0 | 62.6 | 54.5 | 39.4 | 55.9 | 63.6
  EOT | 56.4 | 57.9 | 54.1 | 34.2 | 56.4 | 64.7

22. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score < 2.6 at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. If the DAS28 score was less than 2.6, the participant was considered to be in DAS28 remission.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 2.4 | 12.8 | 19.3
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 10.4, 95% CI 2-sided [4.3 to 16.5] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 16.9, 95% CI 2-sided [10.0 to 23.9] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

23. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score < 2.6 Through Week 52
Description: as for outcome 22
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: FAS. Here, Number of participants analyzed signifies participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 172 | 171 | 37 | 38 | 39 | 34
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170 | 37 | 38 | 39 | 34
  Week 4 | 4.1 | 5.9 | 0.0 | 0.0 | 2.6 | 0.0
  Week 8: number analyzed (Participants) | 168 | 166 | 37 | 38 | 39 | 34
  Week 8 | 8.9 | 12.7 | 0.0 | 0.0 | 2.6 | 2.9
  Week 12: number analyzed (Participants) | 168 | 166 | 37 | 37 | 39 | 34
  Week 12 | 13.1 | 19.9 | 0.0 | 0.0 | 5.1 | 5.9
  Week 16: number analyzed (Participants) | 166 | 165 | 37 | 37 | 39 | 34
  Week 16 | 18.1 | 24.2 | 0.0 | 10.8 | 10.3 | 2.9
  Week 20: number analyzed (Participants) | 164 | 163 | 37 | 37 | 39 | 34
  Week 20 | 22.6 | 33.1 | 5.4 | 10.8 | 7.7 | 5.9
  Week 24: number analyzed (Participants) | 161 | 160 | 36 | 36 | 39 | 34
  Week 24 | 28.0 | 31.3 | 5.6 | 27.8 | 12.8 | 5.9
  Week 28: number analyzed (Participants) | 158 | 159 | 36 | 36 | 39 | 34
  Week 28 | 30.4 | 32.1 | 11.1 | 22.2 | 12.8 | 8.8
  Week 32: number analyzed (Participants) | 157 | 155 | 36 | 36 | 39 | 34
  Week 32 | 33.8 | 41.3 | 22.2 | 30.6 | 15.4 | 26.5
  Week 36: number analyzed (Participants) | 153 | 155 | 36 | 35 | 37 | 33
  Week 36 | 32.7 | 40.0 | 13.9 | 37.1 | 13.5 | 24.2
  Week 40: number analyzed (Participants) | 151 | 152 | 35 | 34 | 36 | 33
  Week 40 | 37.1 | 36.2 | 20.0 | 35.3 | 22.2 | 30.3
  Week 44: number analyzed (Participants) | 147 | 153 | 34 | 33 | 36 | 33
  Week 44 | 34.0 | 37.3 | 17.6 | 24.2 | 25.0 | 30.3
  Week 48: number analyzed (Participants) | 147 | 151 | 33 | 33 | 35 | 33
  Week 48 | 33.3 | 40.4 | 21.2 | 39.4 | 34.3 | 36.4
  Week 52: number analyzed (Participants) | 145 | 147 | 33 | 33 | 34 | 33
  Week 52 | 38.6 | 42.9 | 27.3 | 36.4 | 26.5 | 39.4
  EOT | 34.9 | 38.6 | 24.3 | 31.6 | 25.6 | 41.2

24. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score <= 3.2 at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. DAS28 score of less than or equal to 3.2 was considered to be low disease activity.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 12.4 | 47.1 | 57.9
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 34.7, 95% CI 2-sided [25.1 to 44.2] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 45.5, 95% CI 2-sided [36.0 to 55.0] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

25. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score <= 3.2 Through Week 52
Description: as for outcome 24
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 22.4 | 24.1
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 36.3 | 44.0
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 47.0 | 59.6
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 55.4 | 63.6
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 62.2 | 69.9
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 67.1 | 71.9
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 67.7 | 76.7
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 65.6 | 70.3
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 69.3 | 73.5
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | 76.3 | 80.4
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | 70.5 | 82.4
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | 73.6 | 78.8
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 71.7 | 77.6
  EOT | 66.9 | 71.3

26. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score <= 3.2 at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. DAS28 score of less than or equal to 3.2 was considered to be low disease activity.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 4.7 | 25.0 | 36.3
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 20.3, 95% CI 2-sided [12.5 to 28.1] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 31.5, 95% CI 2-sided [23.1 to 40.0] — C.I. was based on normal approximation to the binomial distribution (continuity corrected)

27. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score <= 3.2 Through Week 52
Description: as for outcome 26
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 10.6 | 12.9
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 17.9 | 29.5
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 25.6 | 37.3
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 34.9 | 44.2
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 44.5 | 48.5
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 52.2 | 57.5
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 49.4 | 56.0
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 52.2 | 56.1
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 53.6 | 56.8
  Week 40: number analyzed (Participants) | 151 | 152
  Week 40 | 58.3 | 60.5
  Week 44: number analyzed (Participants) | 147 | 153
  Week 44 | 53.7 | 60.8
  Week 48: number analyzed (Participants) | 147 | 151
  Week 48 | 55.8 | 62.9
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 55.2 | 60.5
  EOT | 50.6 | 57.3

28. Secondary Outcome: Change From Baseline in CRP at Week 12
Description: Higher CRP indicates greater disease activity.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
mg/dL | -0.001 (2.038) | -1.499 (1.855) | -1.421 (2.182)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: CRP Change = Treatment + Baseline CRP; LS Mean Difference = -1.597, 95% CI 2-sided [-1.948 to -1.247], Standard Error of Mean 0.178
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; LS Mean Difference = -1.458, 95% CI 2-sided [-1.852 to -1.065], Standard Error of Mean 0.200

29. Secondary Outcome: Change From Baseline in CRP Through Week 52
Description: Higher CRP indicates greater disease activity.
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
mg/dL
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -1.055 (1.539) | -1.411 (1.652)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -1.207 (1.839) | -1.569 (1.769)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -1.532 (1.849) | -1.458 (2.170)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -1.666 (1.828) | -1.513 (2.083)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -1.660 (2.050) | -1.660 (2.179)
  Week 24: number analyzed (Participants) | 161 | 161
  Week 24 | -1.774 (2.022) | -1.721 (2.055)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -1.803 (2.150) | -1.721 (2.151)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -1.844 (2.214) | -1.640 (2.411)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -1.832 (2.005) | -1.696 (2.500)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -1.833 (2.156) | -1.716 (2.329)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -1.815 (1.948) | -1.725 (2.324)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -1.771 (2.189) | -1.751 (2.338)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -1.841 (2.102) | -1.912 (1.992)
  EOT | -1.545 (2.315) | -1.629 (2.386)

30. Secondary Outcome: Change From Baseline in ESR at Week 12
Description: Higher ESR indicates greater disease activity.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
mm/h | -2.42 (19.71) | -18.90 (19.85) | -22.17 (22.79)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: ESR Change = Treatment + Baseline ESR; LS Mean Difference = -17.89, 95% CI 2-sided [-21.61 to -14.17], Standard Error of Mean 1.89
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: ESR Change = Treatment + Baseline ESR; LS Mean Difference = -20.61, 95% CI 2-sided [-24.67 to -16.56], Standard Error of Mean 2.06

31. Secondary Outcome: Change From Baseline in ESR Through Week 52
Description: Higher ESR indicates greater disease activity.
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 170
mm/h
  Week 4: number analyzed (Participants) | 170 | 169
  Week 4 | -11.09 (14.34) | -16.59 (16.68)
  Week 8: number analyzed (Participants) | 168 | 165
  Week 8 | -14.96 (18.73) | -21.10 (20.37)
  Week 12: number analyzed (Participants) | 168 | 165
  Week 12 | -19.14 (19.81) | -22.92 (22.66)
  Week 16: number analyzed (Participants) | 166 | 164
  Week 16 | -21.42 (19.70) | -24.29 (23.14)
  Week 20: number analyzed (Participants) | 164 | 162
  Week 20 | -23.22 (20.78) | -26.20 (24.12)
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | -25.35 (22.48) | -27.36 (23.23)
  Week 28: number analyzed (Participants) | 158 | 158
  Week 28 | -26.03 (23.70) | -27.88 (24.27)
  Week 32: number analyzed (Participants) | 157 | 154
  Week 32 | -26.92 (23.85) | -27.21 (24.92)
  Week 36: number analyzed (Participants) | 153 | 154
  Week 36 | -25.95 (22.68) | -27.25 (25.10)
  Week 40: number analyzed (Participants) | 152 | 151
  Week 40 | -25.86 (24.41) | -27.74 (24.86)
  Week 44: number analyzed (Participants) | 149 | 152
  Week 44 | -27.13 (22.73) | -27.99 (23.93)
  Week 48: number analyzed (Participants) | 148 | 150
  Week 48 | -25.63 (24.72) | -27.83 (23.29)
  Week 52: number analyzed (Participants) | 145 | 146
  Week 52 | -26.86 (23.60) | -29.12 (23.28)
  EOT | -24.00 (24.49) | -26.11 (25.22)

32. Secondary Outcome: Percentage of Participants With a European League Against Rheumatism (EULAR) Good Response Using DAS28-CRP at Week 12
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good response have been reported in this outcome measure.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 10.1 | 43.0 | 55.6
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 33.0, 95% CI 2-sided [23.7 to 42.2] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 45.5, 95% CI 2-sided [36.2 to 54.8] — CI was based on normal approximation to the binomial distribution (continuity corrected)

33. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-CRP Through Week 52
Description: as for outcome 32
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 19.4 | 21.8
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 30.4 | 41.0
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 42.9 | 57.2
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 51.8 | 60.0
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 59.1 | 68.1
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 65.2 | 70.0
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 63.3 | 74.2
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 63.1 | 69.0
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 67.3 | 72.9
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | 73.7 | 79.1
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | 65.8 | 81.0
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | 71.6 | 78.1
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 69.0 | 76.9
  EOT | 64.5 | 70.8

34. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-CRP at Week 12
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good or moderate response have been reported in this outcome measure.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 35.5 | 77.9 | 84.8
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 42.4, 95% CI 2-sided [32.3 to 52.5] — CI was based on normal approximation to the binomial distribution (continuity corrected
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 49.3, 95% CI 2-sided [39.7 to 58.9] — CI was based on normal approximation to the binomial distribution (continuity corrected

35. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-CRP Through Week 52
Description: as for outcome 34
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 67.1 | 77.1
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 73.8 | 80.1
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 78.6 | 85.5
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 84.3 | 89.1
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 86.6 | 91.4
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 89.4 | 95.6
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 91.1 | 93.7
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 93.0 | 94.2
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 94.8 | 95.5
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | 92.8 | 96.1
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | 95.3 | 94.1
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | 95.3 | 97.4
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 95.2 | 94.6
  EOT | 88.4 | 92.4

36. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-ESR at Week 12
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good response have been reported in the outcome measure.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 4.1 | 23.8 | 34.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; No multiplicity adjustment; Percent Difference = 19.7, 95% CI 2-sided [12.1 to 27.3] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 30.4, 95% CI 2-sided [22.0 to 38.7] — CI was based on normal approximation to the binomial distribution (continuity corrected)

37. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-ESR Through Week 52
Description: as for outcome 32
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 7.6 | 12.4
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 16.1 | 28.3
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 24.4 | 35.5
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 34.3 | 43.6
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 43.3 | 46.0
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 51.6 | 55.6
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 48.1 | 54.1
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 51.0 | 54.8
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 53.6 | 54.8
  Week 40: number analyzed (Participants) | 151 | 152
  Week 40 | 57.6 | 58.6
  Week 44: number analyzed (Participants) | 147 | 153
  Week 44 | 52.4 | 59.5
  Week 48: number analyzed (Participants) | 147 | 151
  Week 48 | 53.7 | 60.9
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 53.8 | 59.2
  EOT | 49.4 | 56.1

38. Secondary Outcome: Percentage of Participants With a EULAR Good or Moderate Response Using DAS28-ESR at Week 12
Description: as for outcome 34
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 32.0 | 74.4 | 78.9
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 42.5, 95% CI 2-sided [32.3 to 52.6] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 47.0, 95% CI 2-sided [37.1 to 56.9] — CI was based on normal approximation to the binomial distribution (continuity corrected)

39. Secondary Outcome: Percentage of Participants With a EULAR Good or Moderate Response Using DAS28-ESR Through Week 52
Description: as for outcome 34
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 55.9 | 68.2
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 72.0 | 76.5
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 75.0 | 80.1
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 80.7 | 87.9
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 82.3 | 92.0
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 87.6 | 91.9
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 88.0 | 91.2
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 90.4 | 92.9
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 94.1 | 94.8
  Week 40: number analyzed (Participants) | 151 | 152
  Week 40 | 92.7 | 94.1
  Week 44: number analyzed (Participants) | 147 | 153
  Week 44 | 96.6 | 94.1
  Week 48: number analyzed (Participants) | 147 | 151
  Week 48 | 94.6 | 95.4
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 93.8 | 94.6
  EOT | 86.0 | 90.6

40. Secondary Outcome: Percentage of Participants Achieving ACR / EULAR Remission at Week 12
Description: ACR/EULAR Remission was defined as TJC (68 joints) ≤ 1, SJC (66 joints) ≤1, CRP ≤1 mg/dL, and participant's global assessment of arthritis ≤ 1 cm (on a visual analog scale (VAS) of 0 - 100 mm).
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 0.6 | 5.8 | 9.9
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.011, Fisher Exact — No multiplicity adjustment; Percent Difference = 5.2, 95% CI 2-sided [1.0 to 9.5] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 9.3, 95% CI 2-sided [4.1 to 14.6] — CI was based on normal approximation to the binomial distribution (continuity corrected)

41. Secondary Outcome: Percentage of Participants Achieving ACR / EULAR Remission Through Week 52
Description: as for outcome 40
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 1.2 | 1.2
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 1.2 | 3.6
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 6.0 | 10.2
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 9.0 | 12.1
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 11.0 | 14.1
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 11.8 | 18.1
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 14.6 | 20.1
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 17.2 | 25.8
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 17.0 | 27.7
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | 19.1 | 20.9
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | 16.1 | 20.3
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | 17.6 | 21.2
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 21.4 | 26.5
  EOT | 19.2 | 23.4

42. Secondary Outcome: Percentage of Participants Achieving Simplified Disease Activity Index (SDAI) Remission <=3.3 at Week 12
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to description. SDAI = TJC + SJC + SGA + PGA + CRP. SDAI Remission was defined as SDAI score ≤ 3.3.
Time Frame: Week 12/ET
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 169 | 172 | 171
percentage of participants | 0.6 | 7.0 | 14.0
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority — No multiplicity adjustment; p = 0.003, Fisher Exact; Percent Difference = 6.4, 95% CI 2-sided [1.8 to 11.0] — CI was based on normal approximation to the binomial distribution (continuity corrected)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — No multiplicity adjustment; Percent Difference = 13.4, 95% CI 2-sided [7.5 to 19.4] — CI was based on normal approximation to the binomial distribution (continuity corrected)

43. Secondary Outcome: Percentage of Participants Achieving SDAI Remission Score <=3.3 Through Week 52
Description: as for outcome 42
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
percentage of participants
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 1.2 | 2.4
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 3.0 | 8.4
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 7.1 | 14.5
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | 14.5 | 18.2
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | 18.3 | 20.9
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | 20.5 | 22.5
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 22.2 | 23.3
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | 25.5 | 28.4
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | 24.2 | 32.9
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | 31.6 | 28.8
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | 27.5 | 30.1
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | 25.7 | 32.5
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 30.3 | 39.5
  EOT | 28.5 | 35.1

44. Secondary Outcome: Change From Baseline in SDAI Score at Week 12
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to description: SDAI = TJC + SJC + SGA + PGA + CRP. The SDAI score ranges from 0 to approximately 86. Higher SDAI indicates greater disease activity.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -4.90 (12.32) | -15.66 (12.69) | -19.57 (13.53)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SDAI Change = Treatment + Baseline SDAI; LS Mean Difference = -11.22, 95% CI 2-sided [-13.84 to -8.60], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SDAI Change = Treatment + Baseline SDAI; LS Mean Difference = -14.67, 95% CI 2-sided [-17.35 to -11.98], Standard Error of Mean 1.36

45. Secondary Outcome: Change From Baseline in SDAI Score Through Week 52
Description: as for outcome 44
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -11.02 (8.23) | -13.79 (10.43)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -14.60 (10.40) | -18.36 (11.76)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -15.94 (12.59) | -20.08 (13.08)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -18.75 (11.58) | -22.21 (12.56)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -20.24 (11.89) | -23.03 (13.26)
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | -21.62 (11.64) | -24.68 (11.52)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -21.89 (11.54) | -24.57 (12.17)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -22.61 (11.15) | -25.38 (11.91)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -22.89 (11.10) | -25.55 (11.74)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -23.55 (11.20) | -26.14 (11.93)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -23.55 (11.17) | -26.44 (12.15)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -23.23 (11.30) | -26.50 (12.12)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -23.67 (11.91) | -26.63 (12.82)
  EOT | -21.48 (13.42) | -24.72 (14.13)

46. Secondary Outcome: Change From Baseline in PGA at Week 12
Description: The investigator assessed the participants' disease activity on a VAS of 0-100 mm on the physician assessment table. Higher PGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -11.88 (21.46) | -28.83 (22.21) | -35.96 (25.00)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: PGA (100 mm VAS) Change = Treatment + Baseline PGA (100 mm VAS); LS Mean difference = -17.67, 95% CI 2-sided [-22.11 to -13.22], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: PGA (100 mm VAS) Change = Treatment + Baseline PGA (100 mm VAS); LS Mean Difference = -24.09, 95% CI [-28.66 to -19.51], Standard Error of Mean 2.33

47. Secondary Outcome: Change From Baseline in PGA Through Week 52
Description: The investigator assessed the participants disease activity on a VAS of 0-100 mm on the physician assessment table. Higher PGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -18.36 (17.10) | -22.94 (19.32)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -25.79 (19.59) | -31.54 (22.43)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -29.07 (22.22) | -36.55 (24.64)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -33.60 (21.27) | -38.86 (23.83)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -36.18 (21.87) | -41.44 (22.71)
  Week 24: number analyzed (Participants) | 161 | 160
  Week 24 | -37.13 (21.71) | -43.67 (21.39)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -38.72 (22.45) | -42.43 (21.27)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -40.04 (20.82) | -43.96 (21.78)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -39.35 (21.25) | -44.37 (21.77)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -41.04 (22.33) | -44.32 (21.54)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -41.47 (22.73) | -46.00 (21.60)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -41.55 (23.23) | -45.84 (21.83)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -41.49 (23.75) | -45.46 (23.75)
  EOT | -38.41 (25.07) | -43.33 (24.31)

48. Secondary Outcome: Change From Baseline in SGA at Week 12
Description: The participant assessed his/her own disease activity on a VAS of 0-100 mm on the questionnaire form. Higher SGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -7.11 (23.05) | -21.09 (23.63) | -26.57 (25.43)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SGA (100 mm VAS) Change = Treatment + Baseline SGA (100 mm VAS); LS Mean Difference = -16.64, 95% CI 2-sided [-21.09 to -12.19], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SGA (100 mm VAS) Change = Treatment + Baseline SGA (100 mm VAS); LS Mean difference = -20.34, 95% CI 2-sided [-25.07 to -15.61], Standard Error of Mean 2.40

49. Secondary Outcome: Change From Baseline in SGA Through Week 52
Description: as for outcome 48
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -13.80 (19.47) | -17.59 (20.25)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -19.11 (23.22) | -24.97 (22.65)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -21.59 (23.43) | -27.40 (24.84)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -25.20 (24.41) | -30.14 (24.29)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -26.94 (25.49) | -31.20 (25.39)
  Week 24: number analyzed (Participants) | 161 | 161
  Week 24 | -29.00 (25.51) | -32.79 (25.68)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -30.04 (24.96) | -34.25 (25.01)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -31.92 (24.99) | -33.46 (24.28)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -32.38 (25.34) | -34.01 (23.83)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -32.80 (25.85) | -34.24 (23.85)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -33.49 (25.86) | -35.31 (25.23)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -33.69 (26.18) | -35.33 (23.77)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -33.18 (27.83) | -36.16 (25.27)
  EOT | -29.34 (28.78) | -34.05 (26.60)

50. Secondary Outcome: Change From Baseline in SGAP at Week 12
Description: The participant assessed his/her own pain severity on a visual analog scale (VAS) of 0-100 mm on the questionnaire form. Higher SGA of pain (100 mm VAS) scores indicated greater activity pain.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -6.64 (25.22) | -21.09 (27.04) | -26.87 (26.65)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SGAP (100 mm VAS) Change = Treatment + Baseline SGAP (100 mm VAS); LS Mean Difference = -17.19, 95% CI 2-sided [-22.00 to -12.38], Standard Error of Mean 2.44
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SGAP (100 mm VAS) Change = Treatment + Baseline SGAP (100 mm VAS); LS Mean difference = -20.89, 95% CI 2-sided [-25.80 to -15.98], Standard Error of Mean 2.50

51. Secondary Outcome: Change From Baseline in SGAP Through Week 52
Description: as for outcome 50
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -12.94 (20.75) | -16.18 (22.06)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -19.10 (25.81) | -24.98 (23.68)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -21.27 (27.03) | -27.81 (26.13)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -24.03 (26.09) | -28.42 (26.88)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -25.57 (28.52) | -30.63 (26.68)
  Week 24: number analyzed (Participants) | 161 | 161
  Week 24 | -27.34 (27.54) | -32.72 (26.04)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -28.54 (27.24) | -34.18 (25.89)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -31.32 (25.76) | -33.74 (25.44)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -31.95 (26.17) | -32.66 (26.25)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -32.17 (26.81) | -34.07 (25.22)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -32.73 (26.67) | -34.88 (25.27)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -33.60 (25.87) | -35.07 (25.05)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -33.34 (26.98) | -35.00 (27.37)
  EOT | -28.94 (28.63) | -32.68 (28.48)

52. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Participants who discontinued due to lack of efficacy have been reported.
Time Frame: Up to week 52
Population: FAS.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo / Peficitinib 100 mg: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 12 or 28 were switched to receive 100 mg tablet of peficitinib orally once daily in combination with MTX from week 12 or 28 to week 52.
- Placebo / Peficitinib 150 mg: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 12 or 28 were switched to receive 150 mg tablet of peficitinib orally once daily in combination with MTX from week 12 or 28 to week 52.
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg
Number analyzed (Participants) | 175 | 174 | 85 | 85
Participants | 10 | 6 | 3 | 9

53. Secondary Outcome: Change From Baseline in HAQ-DI at Week 12
Description: Participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | 0.01 (0.47) | -0.22 (0.44) | -0.37 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: HAQ-DI Change = Treatment + Baseline HAQ-DI; LS Mean Difference = -0.27, 95% CI 2-sided [-0.36 to -0.17], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: HAQ-DI Change = Treatment + Baseline HAQ-DI; LS Mean Difference = -0.39, 95% CI 2-sided [-0.48 to -0.29], Standard Error of Mean 0.05

54. Secondary Outcome: Change From Baseline in HAQ-DI Through Week 52
Description: as for outcome 53
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | -0.08 (0.30) | -0.21 (0.36)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | -0.18 (0.41) | -0.32 (0.42)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | -0.23 (0.44) | -0.38 (0.47)
  Week 16: number analyzed (Participants) | 166 | 165
  Week 16 | -0.30 (0.46) | -0.41 (0.51)
  Week 20: number analyzed (Participants) | 164 | 163
  Week 20 | -0.33 (0.48) | -0.47 (0.53)
  Week 24: number analyzed (Participants) | 161 | 161
  Week 24 | -0.36 (0.50) | -0.48 (0.52)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | -0.36 (0.51) | -0.51 (0.52)
  Week 32: number analyzed (Participants) | 157 | 155
  Week 32 | -0.37 (0.51) | -0.53 (0.54)
  Week 36: number analyzed (Participants) | 153 | 155
  Week 36 | -0.39 (0.50) | -0.53 (0.52)
  Week 40: number analyzed (Participants) | 152 | 153
  Week 40 | -0.42 (0.50) | -0.56 (0.52)
  Week 44: number analyzed (Participants) | 149 | 153
  Week 44 | -0.45 (0.50) | -0.54 (0.53)
  Week 48: number analyzed (Participants) | 148 | 151
  Week 48 | -0.44 (0.49) | -0.56 (0.53)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | -0.43 (0.51) | -0.56 (0.54)
  EOT | -0.36 (0.55) | -0.51 (0.56)

55. Secondary Outcome: Change From Baseline in Short Form Health Survey - 36 Questions, Version 2 (SF-36v2) Physical Component Summary Score at Week 12
Description: The SF-36v2 was scored for the 8 subscales (each range: 0-100 scale): 1. physical functioning, 2. role physical, 3. bodily pain, 4. general health, 5. vitality, 6. social functioning, 7. role-emotional, and 8. mental health. Physical Component Summary Score, Mental Component Summary Score and Roll/Social Component Summary Score were calculated based on the 2007 General Japanese Population Means and Standard Deviations and coefficient. Component summary measures had means of 50 in 2007 General Japanese Population and deviation was expressed by the scale of 10. Higher score indicated better health state.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | 0.57 (12.08) | 6.60 (11.06) | 9.02 (11.54)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 6.41, 95% CI 2-sided [4.09 to 8.74], Standard Error of Mean 1.18
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 8.61, 95% CI 2-sided [6.36 to 10.86], Standard Error of Mean 1.14

56. Secondary Outcome: Change From Baseline in SF-36v2 Physical Component Summary Score Through Week 52
Description: as for outcome 55
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 3.84 (8.91) | 5.77 (11.05)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 4.92 (10.82) | 7.91 (11.88)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 6.68 (11.08) | 9.32 (11.55)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 9.89 (11.86) | 12.44 (11.88)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 11.27 (12.05) | 12.45 (12.45)
  EOT | 9.92 (12.81) | 11.51 (12.77)

57. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Summary Score at Week 12
Description: as for outcome 55
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | 1.07 (8.27) | 3.28 (7.47) | 2.50 (8.44)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 2.70, 95% CI 2-sided [1.21 to 4.18], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.036, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 1.65, 95% CI 2-sided [0.11 to 3.19], Standard Error of Mean 0.78

58. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Summary Score Through Week 52
Description: as for outcome 55
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 1.45 (7.02) | 1.33 (7.93)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 2.72 (7.39) | 2.44 (8.47)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 3.44 (7.47) | 2.67 (8.23)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 3.06 (8.55) | 3.12 (8.20)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 2.62 (9.10) | 1.85 (8.71)
  EOT | 2.21 (8.89) | 1.67 (8.90)

59. Secondary Outcome: Change From Baseline in SF-36v2 Role/Social Component Summary Score at Week 12
Description: as for outcome 55
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 172 | 171
units on a scale | -0.09 (16.69) | 2.30 (13.92) | 3.90 (13.35)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.099, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 2.29, 95% CI 2-sided [-0.44 to 5.02], Standard Error of Mean 1.39
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.002, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: SF36-v2 Change = Treatment + Baseline SF36-v2; LS Mean Difference = 4.22, 95% CI 2-sided [1.53 to 6.91], Standard Error of Mean 1.37

60. Secondary Outcome: Change From Baseline in SF-36v2 Role/Social Component Summary Score Through Week 52
Description: as for outcome 55
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 172 | 171
units on a scale
  Week 4: number analyzed (Participants) | 170 | 170
  Week 4 | 1.41 (11.51) | 1.70 (11.44)
  Week 8: number analyzed (Participants) | 168 | 166
  Week 8 | 2.50 (13.79) | 3.30 (13.43)
  Week 12: number analyzed (Participants) | 168 | 166
  Week 12 | 2.32 (14.05) | 3.92 (13.31)
  Week 28: number analyzed (Participants) | 158 | 159
  Week 28 | 4.06 (14.92) | 4.81 (13.83)
  Week 52: number analyzed (Participants) | 145 | 147
  Week 52 | 4.30 (15.31) | 7.17 (14.05)
  EOT | 3.49 (14.85) | 5.88 (14.31)

61. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Percent Work Time Missed at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent work time missed due to problem was calculated as Q2/(Q2+Q4). Negative values indicate improvement from baseline.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent work time missed
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 98 | 82 | 95
percent work time missed | -0.82 (17.77) | 0.36 (18.15) | -1.46 (15.26)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.879, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -0.37, 95% CI 2-sided [-5.16 to 4.42], Standard Error of Mean 2.43
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.377, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -1.81, 95% CI 2-sided [-5.86 to 2.23], Standard Error of Mean 2.05

62. Secondary Outcome: Change From Baseline in WPAI Percent Work Time Missed Through Week 52
Description: as for outcome 61
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent work time missed
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 82 | 95
percent work time missed
  Week 4: number analyzed (Participants) | 80 | 91
  Week 4 | -0.90 (16.50) | 0.02 (16.53)
  Week 8: number analyzed (Participants) | 77 | 89
  Week 8 | -1.48 (15.72) | -1.73 (16.59)
  Week 12: number analyzed (Participants) | 77 | 89
  Week 12 | -0.70 (14.69) | -1.97 (12.14)
  Week 28: number analyzed (Participants) | 70 | 86
  Week 28 | -0.58 (19.15) | -3.49 (13.77)
  Week 52: number analyzed (Participants) | 64 | 79
  Week 52 | -1.93 (12.14) | -1.66 (18.74)
  EOT | -1.76 (14.68) | -1.66 (20.31)

63. Secondary Outcome: Change From Baseline in WPAI Percent Impairment While Working at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent impairment while working due to problem was calculated as Q5/10. Negative values indicate improvement from baseline.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent work impairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 95 | 82 | 94
percent work impairment | -2.42 (27.78) | -11.71 (25.62) | -15.96 (28.30)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.007, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -9.63, 95% CI 2-sided [-16.54 to -2.73], Standard Error of Mean 3.50
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -14.17, 95% CI 2-sided [-21.24 to -7.10], Standard Error of Mean 3.58

64. Secondary Outcome: Change From Baseline in WPAI Percent Impairment While Working Through Week 52
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent impairment while working due to problem was calculates as Q5/10. Negative values indicate improvement from baseline.
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent work impairment
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 83 | 94
percent work impairment
  Week 4: number analyzed (Participants) | 80 | 90
  Week 4 | -10.00 (22.39) | -6.56 (29.31)
  Week 8: number analyzed (Participants) | 76 | 88
  Week 8 | -12.50 (24.93) | -13.98 (26.37)
  Week 12: number analyzed (Participants) | 76 | 89
  Week 12 | -11.97 (26.33) | -16.29 (27.77)
  Week 28: number analyzed (Participants) | 68 | 86
  Week 28 | -20.00 (25.27) | -21.40 (25.21)
  Week 52: number analyzed (Participants) | 64 | 79
  Week 52 | -22.97 (29.90) | -22.41 (28.16)
  EOT | -17.35 (29.10) | -20.43 (28.85)

65. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent overall work impairment due to problem was calculated as Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)]. Negative values indicate improvement from baseline.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 95 | 81 | 94
percent overall work impairment | -2.75 (28.56) | -11.58 (26.22) | -16.91 (29.23)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.010, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -9.43, 95% CI 2-sided [-16.60 to -2.25], Standard Error of Mean 3.63
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -14.61, 95% CI 2-sided [-21.92 to -7.31], Standard Error of Mean 3.70

66. Secondary Outcome: Change From Baseline in WPAI Percent Overall Work Impairment Through Week 52
Description: as for outcome 65
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 82 | 94
percent overall work impairment
  Week 4: number analyzed (Participants) | 79 | 90
  Week 4 | -10.61 (22.36) | -7.51 (30.12)
  Week 8: number analyzed (Participants) | 76 | 88
  Week 8 | -13.13 (25.07) | -14.67 (26.94)
  Week 12: number analyzed (Participants) | 76 | 89
  Week 12 | -12.15 (26.81) | -17.15 (28.94)
  Week 28: number analyzed (Participants) | 68 | 86
  Week 28 | -20.76 (25.78) | -22.49 (26.69)
  Week 52: number analyzed (Participants) | 64 | 79
  Week 52 | -22.48 (30.96) | -23.40 (29.54)
  EOT | -17.43 (30.01) | -21.59 (29.88)

67. Secondary Outcome: Change From Baseline in WPAI Percent Activity Impairment at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent activity impairment due to problem was calculated as Q6/10. Negative values indicate improvement from baseline.
Time Frame: Baseline and week 12/ET
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent activity impairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 168 | 171 | 170
percent activity impairment | -2.50 (28.19) | -13.98 (27.17) | -19.35 (24.28)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -13.19, 95% CI 2-sided [-18.23 to -8.16], Standard Error of Mean 2.56
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment; Based on ANCOVA Model: WPAI Change = Treatment + Baseline WPAI; LS Mean Difference = -17.61, 95% CI 2-sided [-22.57 to -12.66], Standard Error of Mean 2.52

68. Secondary Outcome: Change From Baseline in WPAI Percent Activity Impairment Through Week 52
Description: as for outcome 67
Time Frame: Baseline, weeks 4, 8, 12, 28, 52 and EOT
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent activity impairment
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 171 | 170
percent activity impairment
  Week 4: number analyzed (Participants) | 169 | 169
  Week 4 | -9.23 (22.81) | -10.65 (22.18)
  Week 8: number analyzed (Participants) | 166 | 164
  Week 8 | -13.07 (26.12) | -17.44 (24.28)
  Week 12: number analyzed (Participants) | 167 | 165
  Week 12 | -13.71 (27.30) | -19.88 (24.32)
  Week 28: number analyzed (Participants) | 157 | 156
  Week 28 | -22.17 (27.25) | -26.99 (24.72)
  Week 52: number analyzed (Participants) | 144 | 146
  Week 52 | -24.10 (31.72) | -26.71 (24.78)
  EOT | -21.58 (31.67) | -23.47 (25.96)

69. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) During the First 12 Weeks
Description: TEAEs were defined as any AE that started or worsened in severity after initial dose of study drug or reference drug through week 52 or withdrawal. TEAEs were summarized using MedDRA (Version 11.1) by System Organ Class (SOC) and Preferred Term (PT). Participants reporting more than 1 AE for a given MedDRA PT were counted only once for that term. Participants reporting more than 1 AE within a SOC were counted only once for the SOC total. Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), AEs were graded as grade 1=mild; grade 2=moderate: grade 3 = severe or medically significant, grade 4 = life threatening, grade 5 = death related to AE.
Time Frame: Week 0 to week 12
Population: SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg
Number analyzed (Participants) | 170 | 174 | 174
Participants
  TEAEs | 84 | 89 | 104
  Drug-related TEAEs | 47 | 57 | 80
  TEAEs leading to death | 0 | 0 | 0
  Serious TEAEs | 4 | 5 | 3
  Drug-related serious TEAEs | 2 | 3 | 3
  ≥ Grade 3 TEAEs | 8 | 9 | 16
  TEAEs leading to permanent discontinuation | 7 | 5 | 5
  Drug-Related AE leading to permanent discont. | 6 | 3 | 5

70. Secondary Outcome: Number of Participants With TEAEs From Week 12 to Week 28
Description: TEAEs were defined as any AE that started or worsened in severity after initial dose of study drug or reference drug through week 52 or withdrawal. TEAEs were summarized using MedDRA (Version 11.1) by SOC and PT. Participants reporting more than 1 AE for a given MedDRA PT were counted only once for that term. Participants reporting more than 1 AE within a SOC were counted only once for the SOC total. Based on NCI-CTCAE, AEs were graded as grade 1=mild; grade 2=moderate: grade 3 = severe or medically significant, grade 4 = life threatening, grade 5 = death related to AE
Time Frame: Week 12 to week 28
Population: SAF. Here, Number of participants analyzed signifies participants with available data.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo / Peficitinib 100 mg at Week 12: Participants who received placebo matching to peficitinib 100 mg orally once daily in combination with MTX until week 12 were switched to receive 100 mg tablet of peficitinib orally once daily in combination with MTX from week 12 to week 52.
- Placebo / Peficitinib 150 mg at Week 12: Participants who received placebo matching to peficitinib 150 mg orally once daily in combination with MTX until week 12 were switched to receive 150 mg tablet of peficitinib orally once daily in combination with MTX from week 12 to week 52.
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12
Number analyzed (Participants) | 82 | 167 | 165 | 37 | 38
Participants
  TEAEs | 50 | 95 | 104 | 21 | 25
  Drug-related TEAEs | 27 | 63 | 72 | 16 | 11
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 2 | 5 | 3 | 0 | 0
  Drug-related serious TEAEs | 2 | 3 | 1 | 0 | 0
  ≥ Grade 3 TEAEs | 5 | 7 | 6 | 1 | 1
  TEAEs leading to permanent discontinuation | 4 | 4 | 1 | 0 | 0
  Drug-Related TEAE leading to permanent dicont. | 3 | 3 | 1 | 0 | 0

71. Secondary Outcome: Number of Participants With TEAEs From Week 28 to Week 52
Description: TEAEs were defined as any AE that started or worsened in severity after initial dose of study drug or reference drug through week 52 or withdrawal. TEAEs were summarized using MedDRA (Version 11.1) by SOC and PT. Participants reporting more than 1 AE for a given MedDRA PT were counted only once for that term. Participants reporting more than 1 AE within a SOC were counted only once for the SOC total. Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), AEs were graded as grade 1=mild; grade 2=moderate: grade 3 = severe or medically significant, grade 4 = life threatening, grade 5 = death related to AE.
Time Frame: Week 28 to week 52, plus 28 days after the week 52 visit for participants who did not enroll in the extension study
Population: SAF. Here, Number of participants analyzed signifies participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg at Week 12 | Placebo / Peficitinib 150 mg at Week 12 | Placebo / Peficitinib 100 mg at Week 28 | Placebo / Peficitinib 150 mg at Week 28
Number analyzed (Participants) | 158 | 158 | 36 | 36 | 39 | 34
Participants
  TEAEs | 114 | 112 | 22 | 27 | 25 | 26
  Drug-related TEAEs | 72 | 74 | 14 | 18 | 17 | 17
  TEAEs leading to death | 0 | 0 | 0 | 0 | 1 | 0
  Serious TEAEs | 10 | 8 | 2 | 1 | 1 | 1
  Drug-related serious TEAEs | 4 | 5 | 2 | 1 | 0 | 1
  ≥ Grade 3 TEAEs | 15 | 15 | 2 | 2 | 2 | 2
  TEAEs leading to permanent discontinuation | 4 | 6 | 3 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to week 12, week 12 to week 28, and week 28 to week 52 plus 28 days after the week 52 visit for participants who did not enroll in the extension study.
Description: SAF.
Groups:
- Week 0 to Week 12: Placebo: Participants received placebo matched to peficitinib orally once daily in combination with MTX until week 12.
- Week 0 to Week 12: Peficitinib 100 mg: Participants received 100 mg tablet of Peficitinib orally once daily in combination with MTX for a period of 12 weeks.
- Week 0 to Week 12: Peficitinib 150 mg: Participants received 150 mg tablet of Peficitinib orally once daily in combination with MTX for a period of 12 weeks.
- Week 12 to Week 28: Placebo: Participants received placebo matched to peficitinib orally once daily in combination with MTX until week 12 and from week 12 to 28.
- Week 12 to Week 28: Peficitinib 100 mg: Participants received 100 mg tablet of Peficitinib orally once daily in combination with MTX until week 12 and from week 12 to 28.
- Week 12 to Week 28: Peficitinib 150 mg: Participants received 150 mg tablet of Peficitinib orally once daily in combination with MTX until week 12 and from week 12 to 28.
- Week 12 to Week 28: Placebo / Peficitinib 100 mg at Week 12: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 12 were switched to receive 100 mg tablet orally once daily in combination with MTX from week 12 to week 28.
- Week 12 to Week 28: Placebo / Peficitinib 150 mg at Week 12: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 12 were switched to receive 150 mg tablet orally once daily in combination with MTX from week 12 to week 28.
- Week 28 to Week 52: Peficitinib 100 mg: Participants received 100 mg tablet of Peficitinib orally once daily in combination with MTX until week 28 and from week 28 to 52.
- Week 28 to Week 52: Peficitinib 150 mg: Participants received 150 mg tablet of Peficitinib orally once daily in combination with MTX until week 28 and from week 28 to 52.
- Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 12: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 12 were switched to receive 100 mg tablet orally once daily in combination with MTX from week 12 to week 52.
- Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 12: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 12 were switched to receive 150 mg tablet orally once daily in combination with MTX from week 12 to week 52.
- Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 28: Participants who received placebo matched to peficitinib 100 mg orally once daily in combination with MTX until week 28 were switched to receive 100 mg tablet orally once daily in combination with MTX from week 28 to week 52.
- Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 28: Participants who received placebo matched to peficitinib 150 mg orally once daily in combination with MTX until week 28 were switched to receive 100 mg tablet orally once daily in combination with MTX from week 28 to week 52.
Arm/Group | Week 0 to Week 12: Placebo | Week 0 to Week 12: Peficitinib 100 mg | Week 0 to Week 12: Peficitinib 150 mg | Week 12 to Week 28: Placebo | Week 12 to Week 28: Peficitinib 100 mg | Week 12 to Week 28: Peficitinib 150 mg | Week 12 to Week 28: Placebo / Peficitinib 100 mg at Week 12 | Week 12 to Week 28: Placebo / Peficitinib 150 mg at Week 12 | Week 28 to Week 52: Peficitinib 100 mg | Week 28 to Week 52: Peficitinib 150 mg | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 12 | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 12 | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 28 | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 28
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/174 | 0/174 | 0/82 | 0/167 | 0/165 | 0/37 | 0/38 | 0/158 | 0/158 | 0/36 | 0/36 | 1/39 | 0/34
Serious Adverse Events (participants affected / at risk) | 4/170 | 5/174 | 3/174 | 2/82 | 5/167 | 3/165 | 0/37 | 0/38 | 10/158 | 8/158 | 2/36 | 1/36 | 1/39 | 1/34
Other Adverse Events (participants affected / at risk) | 42/170 | 54/174 | 61/174 | 26/82 | 56/167 | 60/165 | 14/37 | 11/38 | 63/158 | 73/158 | 16/36 | 22/36 | 15/39 | 20/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Week 0 to Week 12: Placebo (N=170) | Week 0 to Week 12: Peficitinib 100 mg (N=174) | Week 0 to Week 12: Peficitinib 150 mg (N=174) | Week 12 to Week 28: Placebo (N=82) | Week 12 to Week 28: Peficitinib 100 mg (N=167) | Week 12 to Week 28: Peficitinib 150 mg (N=165) | Week 12 to Week 28: Placebo / Peficitinib 100 mg at Week 12 (N=37) | Week 12 to Week 28: Placebo / Peficitinib 150 mg at Week 12 (N=38) | Week 28 to Week 52: Peficitinib 100 mg (N=158) | Week 28 to Week 52: Peficitinib 150 mg (N=158) | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 12 (N=36) | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 12 (N=36) | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 28 (N=39) | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 28 (N=34)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Week 0 to Week 12: Placebo (N=170) | Week 0 to Week 12: Peficitinib 100 mg (N=174) | Week 0 to Week 12: Peficitinib 150 mg (N=174) | Week 12 to Week 28: Placebo (N=82) | Week 12 to Week 28: Peficitinib 100 mg (N=167) | Week 12 to Week 28: Peficitinib 150 mg (N=165) | Week 12 to Week 28: Placebo / Peficitinib 100 mg at Week 12 (N=37) | Week 12 to Week 28: Placebo / Peficitinib 150 mg at Week 12 (N=38) | Week 28 to Week 52: Peficitinib 100 mg (N=158) | Week 28 to Week 52: Peficitinib 150 mg (N=158) | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 12 (N=36) | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 12 (N=36) | Week 28 to Week 52: Placebo / Peficitinib 100 mg at Week 28 (N=39) | Week 28 to Week 52: Placebo / Peficitinib 150 mg at Week 28 (N=34)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (5) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 5 (5) | 6 (6) | 1 (1) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 4 (5) | 1 (2) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (17) | 19 (19) | 16 (16) | 12 (14) | 20 (24) | 19 (22) | 6 (6) | 2 (2) | 25 (27) | 38 (40) | 6 (7) | 6 (6) | 4 (6) | 6 (8)
Pharyngitis (Infections and infestations) | 6 (6) | 3 (3) | 6 (6) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 4 (5) | 5 (5) | 2 (2) | 4 (4) | 2 (4) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 7 (8) | 1 (1) | 1 (1) | 6 (6) | 9 (10) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5) | 2 (2) | 3 (3) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 7 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT02305849/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT02305849/SAP_001.pdf